CLINICAL TRIAL: NCT02837471
Title: Assessing the Feasibility and Usability of a Commercial Medical Grade Pedometer in a Case-managed Home-based Primary and Secondary Cardiovascular Disease Prevention Program for French-speaking Canadians (PiezoRx RCT Study)
Brief Title: Feasibility and Usability of a Pedometer in a Cardiovascular Disease Prevention Program for French-speaking Canadians
Acronym: PiezoRx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: StepsCount Inc (Unknown)
Responsible Party: Principal Investigator, Jennifer Reed, Associate Scientist, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20160491
Record Dates: First submitted 2016-07-01; First posted 2016-07-19 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Cardiovascular Disease
Keywords: Pedometer usability; Usability and feasibility; web application
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group, PiezoRx device (Experimental): Participants will use the PiezoRx pedometer at leisure for 12 weeks, and receive the standard care of the FrancoForme cardiac prevention and rehabilitation program.
  Interventions: Device: PiezoRx medical grade pedometer
- Control group, Standard care (No Intervention): Participants will receive the standard care of the FrancoForme Cardiovascular disease prevention and rehabilitation program.

INTERVENTIONS:
Device: PiezoRx medical grade pedometer — Participants will be asked to freely use the PiezoRx medical grade pedometer for 12 weeks.
  Participants have access to a personal account created online and can record the daily steps count and physical activity.
  Participants will receive the standard care by the FrancoForme Cardiovascular rehabilitation and prevention program
  Arms: Intervention group, PiezoRx device

SUMMARY:
The purpose of this prospective randomized controlled trial (RCT) is to evaluate the feasibility and usability of a commercial pedometer and web application in a case-managed home-based Cardiovascular disease prevention and rehabilitation program for French-speaking Canadians.

DETAILED DESCRIPTION:
A cardiovascular disease (CVD) prevention and rehabilitation program is an evidence-based, standard of care for those who have coronary artery disease or other cardiac conditions; the aim of CVD prevention and rehabilitation program is to minimize disease progression and prevent future cardiovascular events. Behaviour change interventions targeting exercise are effective for improving physical activity levels, but can be intensive and costly. Activity monitors with accompanying web applications may provide a practical compliment to behaviour change interventions as an affordable way to promote and sustain increased physical activity levels, as measured by steps and physical activity levels. To date, no studies have examined the role of a pedometer with accompanying web application on steps and physical activity levels in French-speaking Canadians attending the FrancoForme® cardiac prevention and rehabilitation program at the University of Ottawa Heart Institute. It is also unknown the average daily steps of Canadian Francophone patients. Identifying successful interventions that promote physical activity among CVD prevention and rehabilitation program patients will help to improve their health as well as decrease the risk of first or subsequent cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Francophone (i.e., French-speaking);
* ≥18 years;
* Existing atherosclerotic vascular disease or ≥1 risk factor for CVD (e.g., family history of premature CVD, age [sex dependent], smoking, sedentary lifestyle, diabetes, hypertension, hypercholesterolemia, overweight/obesity);
* Live in the Champlain Region and attending the onsite FrancoForme® intake;
* Have a family physician or nurse practitioner (to order blood tests and titrate medications);
* Patient agrees to sign informed consent.

Exclusion Criteria:

* Unwilling to wear activity monitors;
* Unable to engage in physical activity;
* Does not have access to the internet;
* Unable to attend follow-up visits;
* Unable to provide written, informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-10; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in number of participants who use the PiezoRx device | One year (Baseline to 12 weeks, and baseline to 52 weeks)
  The number of participants who use the device will be defined as the number of participants who create and use the online account during the trial.
Change in frequency of using the PiezoRx device | One year (Baseline to 12 weeks, and baseline to 52 weeks)
  The frequency of usage will be defined as the number of times the participants logon into the online account to upload the steps count and/or physical activity levels.

SECONDARY OUTCOMES:
Changes in moderate to vigorous physical activity time | One year (Baseline to 12 weeks, and baseline to 52 weeks)
  Changes in levels of moderate to vigorous physical activity (in minutes per week) from baseline to follow-ups will be measured by the PiezoRx device.
Number of participants that continue wearing the PiezoRx device beyond the 3 month intervention | One year
  The number of participants who continue wearing the PiezoRx device beyond the 3 month intervention will be defined as the number of participants who continue to use the online account.
Validation of Physical activity questionnaire | One year
  Self-reported physical activity (in minutes/day) using the physical activity questionnaire.
Validation of Physical activity questionnaire | One year
  Self-reported sitting time (in minutes/day) using the physical activity questionnaire.
Analysis of physical activity data (hrs/min) recorded by PiezoRx device and ActiGraph accelerometer and comparing the values. | 7 days
  Data recorded from PiezoRx device and ActiGraph accelerometer will be collected for 7days. Values will be compared to validate the PiezoRx device against the ActiGraph.
Changes in blood pressure | One year (Baseline to 12 weeks, and baseline to 52 weeks)
  Changes in blood pressure (mmHg) from baseline to from baseline to follow-ups
Changes in blood lipids | One year (Baseline to 12 weeks, and baseline to 52 weeks)
  Changes in total cholesterol, HDL, LDL, and Triglycerides (mmol/L) from baseline to follow-ups
Changes in fasting glycosylated hemoglobin | One year (Baseline to 12 weeks, and baseline to 52 weeks)
  Changes in fasting blood HbA1c (%) from baseline to follow-ups
Changes in body weight | One year (Baseline to 12 weeks, and baseline to 52 weeks)
  Changes in body weight (kg) from baseline to follow-ups
Changes in body mass index | One year (Baseline to 12 weeks, and baseline to 52 weeks)
  Changes in BMI (kg/m2) from baseline to follow-ups
Changes in waist circumference | One year (Baseline to 12 weeks, and baseline to 52 weeks)
  Changes in waist circumference (cm) from baseline to follow-ups
Changes in resting heart rate | One year (Baseline to 12 weeks, and baseline to 52 weeks)
  Changes in resting heart rate (bpm) from baseline to follow-ups
Changes in anxiety and depression | One year (Baseline to 12 weeks, and baseline to 52 weeks)
  Changes in measures of anxiety and depression as assessed using the Hospital Anxiety and Depression Scale from baseline to follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Reed, PhD MEd, CS, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (2):
- Canada (2):
  - University of Ottawa Heart Insititue, Ottawa, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: Yes